CLINICAL TRIAL: NCT07292610
Title: Impact of Nut Consumption on Mental Health in Young Adults: a Randomized Controlled Trial
Brief Title: Impact of Nut Consumption on Mental Health in Young Adults
Acronym: NUTS4BRAIN-RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SBPLY/23/180225/000177; SBPLY/23/180225/000177 (Other Grant/Funding Number: Junta de Comunidades de Castilla-La Mancha and co-financed by the European Union)
Record Dates: First submitted 2025-11-13; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Depression Disorder; Anxiety; Mental Health; Stress; Cognition; BDNF; General Wellbeing
Keywords: RCT; Dietary Intervention; Nut consumption; young adults; Randomized controlled trial; Mental Health; Depression; Anxiety; Cognition; University students; Sleep quality; Academic performance; Walnuts; Almonds; Pistachios; Hazelnut; BDNF
MeSH Terms: conditions — Anxiety Disorders; Psychological Well-Being; Depression; Sleep Initiation and Maintenance Disorders | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: A 6-month, randomized, single-blinded, three-arm, dose-response, clinical trial
Masking Description: The allocation sequence will be concealed from the research team until the allocation time. Participants will be informed of their group assignment upon completion of the randomization process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): Usual dietary habits.
  Interventions: Other: control group
- Intervention Group A (Experimental): Nut consumption (walnuts, almonds, pistachios, and hazelnuts mix).
  Interventions: Dietary Supplement: mixed nuts. Group A
- Intervention Group B (Experimental): Nut consumption (walnuts, almonds, pistachios, and hazelnuts mix).
  Interventions: Dietary Supplement: mixed nuts. Group B

INTERVENTIONS:
Dietary Supplement: mixed nuts. Group A — Participants will be instructed to consume a single daily dose of nuts (30 g/day of mixed nuts). Nuts will be provided free of charge for the entire study period (6 moths). The participants will be instructed to incorporate nuts into their regular diet and consume them in any way they prefer.
  Upon completion of the intervention, participants will be instructed to continue their usual dietary and lifestyle habits, without any specific restrictions or incentives directed toward nut consumption. After 6 months have passed since the end of the intervention, all participants will be called for a final session (12 months) in which all data evaluated throughout the study will be collected
  Arms: Intervention Group A
Dietary Supplement: mixed nuts. Group B — Participants will be instructed to consume two daily doses of nuts (60 g/day of mixed nuts). Nuts will be provided free of charge for the entire study period (6 months). The participants will be instructed to incorporate nuts into their regular diet and consume them in any way they prefer.Upon completion of the intervention, participants will be instructed to continue their usual dietary and lifestyle habits, without any specific restrictions or incentives directed toward nut consumption. After 6 months have passed since the end of the intervention, all participants will be called for a final session (12 months) in which all data evaluated throughout the study will be collected
  Arms: Intervention Group B
Other: control group — Participants will be instructed to maintain their regular diet without any specific dietary instructions or intervention.
  Arms: Control Group

SUMMARY:
Nuts have a high nutrient density, and numerous studies have reported their cardiometabolic benefits. Although observational studies in adults have indicated a potential link between nut consumption and improved mental health, there is still insufficient evidence from experimental studies to draw firm conclusions about this association.

DETAILED DESCRIPTION:
Nuts are widely recognized for their high nutrient density and their multiple reported cardiometabolic benefits. They are rich in monounsaturated (MUFAs) and polyunsaturated (PUFAs) fatty acids (including omega-3 alpha-linolenic acid and omega-6 linoleic acid) as well as antioxidants and compounds with anti inflammatory properties. Observational studies in adults have suggested a potential association between nut consumption and improved mental health, including a reduced risk of depression and enhanced mood. However, evidence from experimental studies remains limited and often inconclusive.

Early adulthood (ages 18-24) represents a critical developmental period marked by substantial physical, psychological, and social changes, and it is also a stage during which mental health problems commonly emerge.

The Nuts4Brain-RCT will investigate the impact of a 6-month mixed-nut intervention on mental health symptoms, cognitive functioning, sleep quality, overall well-being, health-related quality of life, and biochemical mediators of brain function and mental health in young adults.

ELIGIBILITY:
Participants must meet all the following criteria to be considered eligible for selection and randomization:

Inclusion Criteria:

* Age: Participants must be between 18 and 25 years old.
* Academic Status: Participants must be enrolled as university students.
* Field of Study: Participants may come from any academic program offered at the Cuenca Campus, including Nursing, Social Work, Education, Fine Arts, Engineering, Journalism, and Teaching.

Participants will be excluded from the study if they have any of the following conditions, based on self-reported information:

Exclusion Criteria:

* Allergies: Known nut allergy.
* Self-reported cardiovascular, metabolic, gastrointestinal or mental health disorder.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Depression | "Day 0", "Month 3", "Month 6", "Month 12"
  Changes in symptoms of depression assessed with the Beck Depression Inventory Version II (BDI-II). Each of the 21 items includes four statements of increasing severity, and a total score (ranging from 0 to 63) is calculated, with higher scores indicating more severe depression.
Anxiety | "Day 0", "Month 3", "Month 6", "Month 12"
  Changes in symptoms of anxiety assessed with The Generalized Anxiety Disorder 7-item (GAD-7). The GAD-7 consists of seven questions asking individuals to rate the frequency and severity of specific anxiety symptoms over the past two weeks.The total score ranges from 0 to 21, calculated by summing the scores of all seven items. A score of 10 or greater is considered a reasonable cut-off point for identifying possible cases of GAD that may require further clinical evaluation
Stress | "Day 0", "Month 3", "Month 6", "Month 12"
  Changes in symptoms of stress assessed with The Perceived Stress Scale (PSS-10). The PSS-10 is a widely used, 10-item self-report questionnaire that measures an individual's perception of stress over the past month. Scoring involves reverse-scoring four positive items and summing all 10. Total scores range from 0 to 40, with higher scores indicating more perceived stress. Scores can be interpreted generally as low (0-13), moderate (14-26), or high (27-40) stress.
Episodic memory | "Day 0", "Month 3", "Month 6", "Month 12"
  The Picture Sequence Memory Test assesses episodic memory by requiring participants to encode and recall the temporal order of a sequence of visually presented everyday events. After presentation, individuals are asked to reconstruct the sequence in its original order, allowing evaluation of visual episodic memory and learning across trials. Test time: 7 minutes. This test is one of the measures included in the NIH Toolbox Cognition Battery, which is administered on an iPad by qualified personnel.
Working memory | "Day 0", "Month 3", "Month 6", "Month 12"
  The List Sorting Working Memory Test (LSWM), part of the NIH Toolbox Cognition Batery, assesses working memory by having individuals recall and sequence visually and auditorily presented stimuli (like animal/food pictures) in size order (smallest to largest). Test time: 7 minutes.
Cognitive flexibility | "Day 0", "Month 3", "Month 6", "Month 12"
  The Dimensional Change Card Sort Test is a standardized measure of cognitive flexibility. Participants are required to sort cards according to different rules (e.g., color or shape) and to adapt their responses when the sorting dimension changes. Test time: 5 minutes.
  This test is one of the tests that will be determined using the NIH Toolbox Cognition Battery, which will be administered on an iPad by qualified personnel.
Processing speed | "Day 0", "Month 3", "Month 6", "Month 12"
  The Pattern Comparison Processing Speed Test is a standardized measure of processing speed. Participants are asked to quickly determine whether two visual patterns are the same or different, emphasizing speed and accuracy of visual perception and decision-making. Test Time: 4 minutes.
  This test is one of the tests that will be determined using the NIH Toolbox Cognition Battery, which will be administered on an iPad by qualified personnel.
Inhibitory control and attention | "Day 0", "Month 3", "Month 6", "Month 12"
  The Flanker Inhibitory Control and Attention Test is a standardized measure of inhibitory control and selective attention, core components of executive function. Participants are required to focus on a central target stimulus while inhibiting interference from surrounding distractor stimuli. Performance reflects the ability to maintain attention, suppress competing responses, and resolve cognitive conflict. Test Time: 3 minutes.
  This test is one of the tests that will be determined using the NIH Toolbox Cognition Battery, which will be administered on an iPad by qualified personnel.
Brain Derived Neurotrophic Factor | "Day 0", "Month 3", "Month 6", "Month 12"
  Changes in blood concentration of brain-derived neurotrophic factor (BDNF), a biochemical mediator of brain functioning

SECONDARY OUTCOMES:
Sleep quality | "Day 0", "Month 3", "Month 6", "Month 12"
  Changes in quality of sleep assessed with the Pittsburgh Sleep Quality Index (PSQI). The PSQI consists of 19 individual self-rated questions (and 5 optional questions for a roommate/bed partner) that are grouped into seven component scores. Each of the seven components is scored on a scale of 0 to 3, where 0 indicates no difficulty and 3 indicates severe difficulty. The scores of these components are summed to produce a global PSQI score, which ranges from 0 to 21. Higher scores indicate poorer sleep quality.
Health-related quality of life (HRQL) | "Day 0", "Month 3", "Month 6", "Month 12"
  Changes in health-related quality of life assessed with the SF12 questionnaire. It consists of 12 questions that cover the same eight health domains as the longer SF-36: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional, and Mental Health.
  The 12 items are used to create two main summary measures through a complex, norm-based scoring algorithm:
  Physical Component Summary (PCS): A single score representing physical health status.
  Mental Component Summary (MCS): A single score representing mental and emotional health status.
  Interpretation of Scores:
  Scores for both PCS and MCS typically range from 0 to 100, where higher scores indicate better health and functioning.
Inflammatory biomarkers | "Day 0", "Month 3", "Month 6", "Month 12"
  Changes in blood inflammatory markers (e.g. hs-CRP) to examine underlying mechanisms
Concentration of vitamins and minerals | "Day 0", "Month 3", "Month 6", "Month 12"
  Changes in blood concentration of specific vitamins and minerals (e.g., vitamins B9, B12, D, iron, and magnesium) to examine underlying mechanisms
Body image | "Day 0", "Month 3", "Month 6", "Month 12"
  Changes in body image perception using The Standard Figural Stimuli (SFS). Measurement Purpose:
  Perceived Body Image: The figure the individual selects as most representative of their current body size.
  Ideal Body Image: The figure the individual would like to have. Body Dissatisfaction: The discrepancy between the perceived image and the ideal image. A larger difference indicates greater body dissatisfaction.
Screen time | "Day 0", "Month 3", "Month 6", "Month 12"
  Screen time will be assessed using an ad hoc questionnaire that records the number of hours of leisure time participants spend watching television, using a mobile phone, using a computer for work-related purposes, or engaging with other electronic devices, both on weekdays and during weekends.
Social media addiction | "Day 0", "Month 3", "Month 6", "Month 12"
  Changes in social media addiction through Social Network Addiction Questionnaire, 6-item version (ARS-6). The scale typically consists of 6 items, with one item representing each of the six components of addiction.
  Response Scale: Responses are typically given on a 5-point Likert scale (e.g., from 1 = Not at all to 5 = Always).
  Scoring: Item responses are summed to obtain a total score, ranging from 6 to 30. Higher scores indicate a greater risk or severity of social media addiction.
Sociodemographic | "Day 0", "Month 3", "Month 6", "Month 12"
  Sociodemographic information such as age, sex, date of birth, country of origin, marital status, housing type, medication use, and family history of mental or cardiovascular disorders.
Drugs consumption | "Day 0", "Month 3", "Month 6", "Month 12"
  Changes in drugs consumption assessed with the Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST). The ASSIST generates substance-specific risk scores that categorize use into low, moderate, or high-risk categories. Higher scores indicate a greater risk of substance-related health and social problems, guiding the type of intervention needed (e.g., brief intervention or referral to specialist treatment).
Adherence to the Mediterranean Diet | "Day 0", "Month 3", "Month 6", "Month 12"
  Changes in adherence to the mediterranean diet assessed with the MEDAS questionnaire.
  Scoring:
  Each item is scored with 1 point if the criteria for adherence to the Mediterranean diet are met, and 0 points if they are not.
  The total score ranges from 0 to 14 points. Higher scores indicate greater adherence to the Mediterranean diet. A common cut-off point of ≥9 is often used to define good adherence to the diet.
Resilience | "Day 0", "Month 3", "Month 6", "Month 12"
  Changes in resilience assessed with the Connor-Davidson Resilience Scale (CD-RISC 10). Each item is rated on a 5-point Likert scale ranging from 0 (not true at all) to 4 (true nearly all the time). The total score is calculated by summing the values of all 10 items. Total scores range from 0 to 40. Higher scores on the CD-RISC 10 indicate greater resilience and a better ability to cope with adversity and bounce back from difficult experiences.
Risk of eating disorders | "Day 0", "Month 3", "Month 6", "Month 12"
  The SCOFF questionnaire (an acronym derived from the initials of its English questions: Sick, Control, One stone, Fat, Food) is a brief and simple, five-question screening tool designed to detect the possible presence of eating disorders (EDs), such as anorexia nervosa and bulimia nervosa. The total score can range from 0 to 5. A score of two or more points is considered a positive screening result and suggests a suspicion of an ED that requires a detailed formal clinical assessment.
Weight | "Day 0", "Month 3", "Month 6", "Month 12"
  Weight in kilograms will be assessed twice using a calibrated digital scale (Scale Seca® 861) with participants barefoot and in light weight clothing.
Height | "Day 0", "Month 3", "Month 6", "Month 12"
  Height will be measured twice with a stadiometer (Wall stadiometer Seca® 222), with participants standing upright, barefoot, and with the sagittal midline aligned to the wall.
Body Mass Index (BMI) | "Day 0", "Month 3", "Month 6", "Month 12"
  BMI will be calculated as weight divided by height squared (kg/m2).
Body fat percentage | "Day 0", "Month 3", "Month 6", "Month 12"
  Body fat percentage will be assessed twice using the bioimpedance analysis system under standardized conditions (morning, fasting, post-void, after 15 minutes rest, barefoot, with controlled temperature and humidity).
Blood pressure | "Day 0", "Month 3", "Month 6", "Month 12"
  Blood pressure will be measured using an automated device (OMRON® M5-I (Omron Healthcare UK Ltd.)). Systolic and diastolic blood pressure will be assessed twice, with a 5-minute interval between measurements. Participants will be seated in a quiet environment, with the right arm semi-flexed at heart level.
Muscular strenght | "Day 0", "Month 3", "Month 6", "Month 12"
  Measured through handgrip strength using a calibrated dynamometer (Digital dynamometer TKK 5401 Grip-D (Takey®, Tokyo, Japan), and standing long jump for lower body strength. Handgrip: Kilograms (kg). Horizontal jump: Centimeters (cm).
Phisical activity | "Day 0", "Month 3", "Month 6", "Month 12"
  Changes in phisical activity assessed with the The International Physical Activity Questionnaire (IPAQ). The data collected with the IPAQ can be reported as a continuous measure (estimation of total energy expenditure in MET-minutes per week) or categorically (classifying individuals into low, moderate, or high physical activity levels):
  Continuous Score: Total energy expenditure is calculated using specific formulas that assign MET (metabolic equivalent) values to each activity type (walking=3.3 METs, moderate=4.0 METs, vigorous=8.0 METs).
  Categorical Score: Participants are classified into three levels of physical activity based on predefined criteria related to the duration, frequency, and intensity of activities.
Lipid profile | "Day 0", "Month 3", "Month 6", "Month 12"
  Changes in blood lipid profile (Cholesterol (Total, HDL-c, LDL-c), triglycerides)) to examine underlying mechanisms.
Glucose levels | "Day 0", "Month 3", "Month 6", "Month 12"
  Changes in blood glucose levels to examine underlying mechanisms.
Hemoglobin A1c (HbA1c) | Day 0", "Month 3", "Month 6", "Month 12"
  Changes in blood HbA1c levels to examine underlying mechanisms.
Adherence verification | "Day 0", "Month 3", "Month 6", "Month 12"
  Adherence to nut consumption intervention measured by blood levels of vitamin E

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Eumann Mesas, PhD, Principal Investigator — Health and Social Research Center
Locations (1):
- Health and Social Research Center. University of Castilla-La Mancha, Cuenca, Cuenca, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data generated in this project will be publicly shared through Zenodo an open-access repository compliant with FAIR (Findable, Accessible, Interoperable, and Reusable) principles.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: These data will remain accessible for a minimum period of five years.
Access Criteria: All data will be securely stored under the responsibility of the project's Principal Investigator, Arthur Eumann Mesas, ensuring compliance with institutional and ethical data protection requirements.